CLINICAL TRIAL: NCT02565251
Title: Volemic Resuscitation in Sepsis and Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Platon Oana, Antal Oana MD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWA00022929
Record Dates: First submitted 2015-09-01; First posted 2015-10-01 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Hemodynamic Instability; Sepsis; Septic Shock
Keywords: sepsis; hemodynamic monitoring; septic shock; volemic resuscitation; fluid resuscitation
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sepsis grup 1 (Experimental): Flotrac/Ev1000 in the first 2 hours and VolumeView/Ev1000 monitoring during the next 4 hours
  Interventions: Device: Flotrac/Ev1000; Device: VolumeView/Ev1000
- Sepsis grup 2 (Experimental): Hemodymanic resuscitation giuded by standard ICU monitorisation (BP, CVP) in the first 2 hours and VolumeView/Ev1000 monitoring during the next 4 hours
  Interventions: Device: Standard ICU monitorisation; Device: VolumeView/Ev1000
- Soc septic grup 1 (Experimental): Flotrac/Ev1000 in the first 2 hours and VolumeView/Ev1000 monitoring during the next 4 hours
  Interventions: Device: Flotrac/Ev1000; Device: VolumeView/Ev1000
- Soc septic grup 2 (Experimental): Hemodymanic resuscitation giuded by standard ICU monitorisation (BP, CVP) in the first 2 hours andVolumeView/Ev1000 monitoring during the next 4 hours
  Interventions: Device: Standard ICU monitorisation; Device: VolumeView/Ev1000

INTERVENTIONS:
Device: Flotrac/Ev1000 — Hemodynamic resusucitation guided by the data obtained from the monitorisation with Flotrac/Ev1000 device in the first two hours
  Arms: Sepsis grup 1; Soc septic grup 1
Device: Standard ICU monitorisation — Hemodynamic resusucitation guided by the data obtained from ICU standard hemodynamic monitoring (BP, CVP) in the first 2 hours
  Arms: Sepsis grup 2; Soc septic grup 2
Device: VolumeView/Ev1000 — Hemodynamic resusucitation guided by the data obtained from the monitorisation with VolumeView/Ev1000 device in the next four hours

SUMMARY:
Severe sepsis and septic shock are among the leading causes of morbidity and mortality in patients admitted in the ICU, being responsible for approximately 200000 deaths/year in the USA and 150000 in Europe. Recognizing the early signs of sepsis and the different stages of this condition may lower the associated morbidity and mortality.

The hemodynamic profile of the septic shock is characterized by the presence of the distributive shock, on which we can add elements from the hypovolemic and cardiogenic shocks.

The objecive of this study is to optimize the volemic resuscitation of the severe septic and of the septic shock patient using two minimally invasive methods of hemdynamic monitoring which both use the same device (Edwards Lifescience). In the same time hemodinamic data will be colected by mesuring the inferior vena cava diameter.

DETAILED DESCRIPTION:
Severe sepsis and septic shock are among the leading causes of morbidity and mortality in patients admitted in the ICU, being responsible for approximately 200000 deaths/year in the USA and 150000 in Europe . Recognizing the early signs of sepsis and the different stages of this condition may lower the associated morbidity and mortality.

The hemodynamic profile of the septic shock is characterized by the presence of the distributive shock, on which we can add elements from the hypovolemic and cardiogenic shocks. The persistence of hypotension after adequate fluid load is the result of low vascular resistance and myocardial dysfunction and calls for certain specific correctional measures.

The diffrent hemodynamic profiles which can be found in the different stages of the septic shock and their dificult clinical identification led to the development of varoius hemodynamic monitoring techniques and devices. These techniques can be classified into invasive and minimally invasive, calibrated and uncalibrated. The major diffrences among these tecniques is the easyness of utilisation and the acuracy of the data obtained.

Inclusion Criteria: severe sepsis and septic shock (acording to the Sepsis Campaign 2013 crieria) patients with medical or surgical pathology which are admitted in the ICU unit in the first six hours after the onset of the severe sepsis/septic shock. The exclusion criteria of the patients are age less then 18 and more then 75, cardiac valvular pathology with hemodynamic importance, cardiac failure NYHA III și IV, primary or secondary pulmonary hypertension with hemodymanic impact with onset before the onset of the septic pathology,severe liver failure (Child-Pugh C), anuric renal failure, pregnant women, patient who refuse blood products adminitration, end-stage cancer.

The objecive of this study is to optimize the volemic resuscitation of the severe septic and of the septic shock patient using two minimally invasive methods of hemdynamic monitoring which both use the same device (Edwards Lifescience). In the same time hemodinamic data will be colected by mesuring the inferior vena cava diameter.

The primary outcome is the adecuacy of tissue perfusion at six hours (urinary output, blood pressure, lactate clearance, skin aspect). The secondary oucomes are duration of cardiovascular failure at the end of the 6 hours resuscitation period/ number of days, duration of respiratory failure (need of mechanical ventilation, number of days), duration of acute renal failure (need of dialysis) at ICU discharge/10/30/60 days, duration of ICU stay and in hospital stay, discharge status at 60 days (not discharged ,discharge to another acute care hospital, discharged to nursing home, discharged home ,other or unknown and all cause mortality at 60 days.

ELIGIBILITY:
Inclusion Criteria: sepsis and septic shock (acording to the Sepsis Campaign 2016 crieria) patients with medical or surgical pathology which are admitted in the ICU unit in the first 12 hours after the onset of the sepsis/septic shock

Exclusion Criteria:

age less then 18 and more then 85 cardiac valvular pathology with hemodynamic importance cardiac failure NYHA IV primary or secondary pulmonary hypertension with hemodymanic impact with onset before the onset of the septic pathology Severe liver failure (Child-Pugh C) Anuric renal failure Pregnant women Patient who refuse blood products adminitration End-stage cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Tissue perfusion at six hours (composite) | six hours
  Tissue perfusion at six hours: urinary output, blood pressure, lactate clearance, skin aspect

SECONDARY OUTCOMES:
Duration of cardiovascular failure | at the end of the 6 hours resuscitation period and one, two, six and twelve days
  need of vasopressor support: at the end of the 6 hours resuscitation period and one, two, six and twelve days
Duration of respiratory failure | respiratory failure at oane day, two days, six days and twelve days
  respiratory failure at oane day, two days, six days and twelve days
Duration of acute renal failure | at 5 days, at 10 days, at 30 days and at 60 days
  Duration of acute renal failure (need of dialysis) at 5 days, at 10 days, at 30 days and at 60 days
Duration of ICU stay and in hospital stay | status at 5 days, at 10 days, at 30 days and at 60 days
  Duration of ICU stay and in hospital stay
Discharge status at 60 days | at 60 days
  Discharge status at 60 days:Not discharged ,Discharge to another acute care hospital,Discharged to nursing home,Discharged home ,Other or unknown
all cause mortality at 60 days | 60 days
  all cause mortality at 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cluj County Emenrgency Hospital, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Result] Lilly CM. The ProCESS trial--a new era of sepsis management. N Engl J Med. 2014 May 1;370(18):1750-1. doi: 10.1056/NEJMe1402564. Epub 2014 Mar 18. No abstract available. PMID 24635774
- [Result] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Result] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Result] Russell JA. Is there a good MAP for septic shock? N Engl J Med. 2014 Apr 24;370(17):1649-51. doi: 10.1056/NEJMe1402066. Epub 2014 Mar 18. No abstract available. PMID 24635771
- [Result] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Result] Bakker J, Nijsten MW, Jansen TC. Clinical use of lactate monitoring in critically ill patients. Ann Intensive Care. 2013 May 10;3(1):12. doi: 10.1186/2110-5820-3-12. PMID 23663301
- [Result] Cecconi M, Arulkumaran N, Kilic J, Ebm C, Rhodes A. Update on hemodynamic monitoring and management in septic patients. Minerva Anestesiol. 2014 Jun;80(6):701-11. Epub 2013 Nov 26. PMID 24280808
- [Result] Cecconi M, Hofer C, Della Rocca G, Grounds RM, Rhodes A. Assessing agreement in cardiac output monitoring validation studies. J Cardiothorac Vasc Anesth. 2010 Aug;24(4):741; author reply 741-2. doi: 10.1053/j.jvca.2009.11.008. Epub 2010 Jan 22. No abstract available. PMID 20096600
- [Result] Monnet X, Anguel N, Naudin B, Jabot J, Richard C, Teboul JL. Arterial pressure-based cardiac output in septic patients: different accuracy of pulse contour and uncalibrated pressure waveform devices. Crit Care. 2010;14(3):R109. doi: 10.1186/cc9058. Epub 2010 Jun 10. PMID 20537159
- [Result] Marque S, Gros A, Chimot L, Gacouin A, Lavoue S, Camus C, Le Tulzo Y. Cardiac output monitoring in septic shock: evaluation of the third-generation Flotrac-Vigileo. J Clin Monit Comput. 2013 Jun;27(3):273-9. doi: 10.1007/s10877-013-9431-z. Epub 2013 Jan 30. PMID 23361128
- [Result] Antonelli M, Levy M, Andrews PJ, Chastre J, Hudson LD, Manthous C, Meduri GU, Moreno RP, Putensen C, Stewart T, Torres A. Hemodynamic monitoring in shock and implications for management. International Consensus Conference, Paris, France, 27-28 April 2006. Intensive Care Med. 2007 Apr;33(4):575-90. doi: 10.1007/s00134-007-0531-4. PMID 17285286